CLINICAL TRIAL: NCT04622371
Title: Effect of Moderate Exercise Versus Breaking Sedentary by Light Exercise on Patients With Type 2 Diabetes Mellitus
Brief Title: Physical Therapy for Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Manal k. youssef, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T. REC/012/002607
Record Dates: First submitted 2020-11-04; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus
Keywords: moderate exercises; light exercises; obesity; sedentary behavior
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: 2-arm cluster randomized controlled trial involved 60 patients aged between 35and 60 years divided randomly into two groups. Group 1 received 30 minutes of aerobic exercise at 40-60% of maximum heart rate. Group 2,Treated by walking30 minutes daily divided into 5minutes every 2 hours to break sedentary position for 12 hours daily.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- moderate exercises group (Experimental): Patients received 30 minutes of aerobic exercise at 40-60% of maximum heart rate
  Interventions: Other: Moderate exercises
- Light exercises group (Experimental): Patients treated by walking30 minutes daily divided into 5minutes every 2 hours to break sedentary position for 12 hours daily.
  Interventions: Other: Moderate exercises

INTERVENTIONS:
Other: Moderate exercises — Group 1 received 30 minutes of aerobic exercise at 40-60% of maximum heart rate. Group 2,Treated by walking30 minutes daily divided into 5minutes every 2 hours to break sedentary position for 12 hours daily.
  Other Names: Light exercises

SUMMARY:
Background: The aim of this study to compare the effect of moderate exercises versus light exercises on patients with type 2 diabetes mellitus.

Methods: This 3-month, 2-arm cluster randomized controlled trial involved 60 patients aged between 35and 60 years divided randomly into two groups. Group 1 received 30 minutes of aerobic exercise at 40-60% of maximum heart rate. Group 2,Treated by walking30 minutes daily divided into 5minutes every 2 hours to break sedentary position for 12 hours daily.

Results: At the base line no significant difference were found in both groups in all parameters. After three months of treatment, there is no significant difference in all parameters BMI, p=0.111, waist to hip ratio, p=0.245, 6 minutes' walk, p=0.614, blood glucose, p=0.105 and sf-36, p=0.106. The study approved by ethical committee of faculty of physical therapy, Cairo University REC/012/002607.

Conclusion: Light exercise has the same effect on blood glucose as moderate exercise, so just walking for 5 minutes every 2 hours can be useful for patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
78 patients have been chosen from department of internal medicine, Cairo university hospitals, Egypt. 8 patients were excluded because 3 have chronic renal failure, 3 have cardiopulmonary diseases and 2 have severe osteoarthritis of knees.

They were divided randomly into two groups, group one will be treated by moderate exercises and group and group 2 will be treated by light exercises.

after division all the procedures were explained to patients.5 patients refused to sign informed consent and excluded from the study.33 patients in group1 and 32 patients in group2.3patients dropped in group1 and excluded from the study and two patients didn't continued the programmed treatment in group 2 and their data removed.

Thirty patients in each group signed an informed consent and complete the treatment program.

ELIGIBILITY:
Inclusion Criteria:

* Type2 diabetes mellitus.
* Age between 35 and 60.
* BMI≥30

Exclusion Criteria:

* Renal failure.
* Cardiopulmonary diseases.
* Lower limb diseases or fracture.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
BMI | 12 week
  Weight divided by square of the height
Waist to hip ratio | 12 weeks
  Circumference of the waist at umbalicus/ circumference of gluteal region
6 minutes walk distance | 12 weeks
  meters walked in 6 minutes
Blood glucose | 12 weeks
  mg/dl
SF-36 | 12 weeks
  degree

CONTACTS AND LOCATIONS:
Overall Officials: Manal K. Youssef, PhD, Principal Investigator — Cairo university, Egypt
Locations (1):
- Manal K. youssef, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared on reasonable request from corresponding author.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 weeks
Access Criteria: Data available on reasonable request from corresponding authors.